CLINICAL TRIAL: NCT05509205
Title: Turkish Adaptation, Validity and Reliability of Pound Satisfaction Scale in Patients With Stroke After Stroke Rehabilitation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Emel Mete, Research Assistant, Istanbul Medeniyet University
Other Study IDs: Pound Satisfaction Scale
Record Dates: First submitted 2022-08-18; First posted 2022-08-22 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Stroke
Keywords: stroke; patient satisfaction; rehabilitation
MeSH Terms: conditions — Stroke; Patient Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with stroke: In this study 130 patients with stroke who are treating with stroke rehabilitation programs, will be included.
  Interventions: Other: Turkish Validity and Reliability of The PSS Scale

INTERVENTIONS:
Other: Turkish Validity and Reliability of The PSS Scale — This study is about validation of the Pound Satisfaction Scale to Turkish. The level of satisfaction with the rehabilitation service and treatment of 130 stroke patients undergoing stroke rehabilitation will be evaluated with the Pound satisfaction scale.

SUMMARY:
The aim of this study is to adapt the Pound Satisfaction Scale (PSS) to Turkish society in stroke patients and to make its validity and reliability in Turkish. The PSS scale developed by Pound et al evaluates the patient's satisfaction with the received rehabilitation program and services received in stroke patients. The PSS scale will be filled in face-to-face with volunteer participants who have received a stroke rehabilitation program and meet the inclusion criteria. 130 participants will be included in the study. In order to assess the concurrent validity of the PSS, the SF-36 (short form) which evaluates the quality of life, and the Patient Satisfaction Scale in Physiotherapy (PSSP) which evaluates patient satisfaction will be used. Scales will be repeated after 15 days to assess test-retest reliability.

DETAILED DESCRIPTION:
The reliability and validity of the scale will begin with language equivalence and cultural adaptation. The scale will be translated from English to Turkish by two people who are fluent in Turkish and English. A single Turkish translation will be obtained from these two Turkish translations with a common opinion. The scale, which has been translated into Turkish, will be translated into English by two other people who are fluent in Turkish and English. The scale translated into English will be compared with the original. If the developer of the scale approves the translation of the scale, participants will be recruited for the study. In the pre-trial phase, a preassessment will be conducted with 15 participants to test the intelligibility of the scale. Based on the results of the pre-test phase, the final version of PSS will be able to be modified. The PSS scale will be filled in face-to-face with volunteer participants who have received a stroke rehabilitation program and meet the inclusion criteria. 130 participants will be included in the study. In order to assess the concurrent validity of the PSS, the SF-36 (short form) which evaluates the quality of life, and the Patient Satisfaction Scale in Physiotherapy (PSSP) which evaluates patient satisfaction will be used. Scales will be repeated after 15 days to assess test-retest reliability.

ELIGIBILITY:
Inclusion Criteria:

* To benefit from Physiotherapy and Rehabilitation services,
* Mini mental state examination (MMSE) score> 24
* Patients with stroke
* Native language being Turkish

Exclusion Criteria:

* Native language not being Turkish
* Patients with motor sequelae from other diseases and insufficient cognitive or educational level to complete the scale
* Mini mental state examination (MMSE) score < 24

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patients who are treating with stroke rehabilitation
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2022-03-02 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-09-10 (Estimated)

PRIMARY OUTCOMES:
Personal Satisfaction | baseline
  Personal Satisfaction will be assessed with Pound Satisfaction Scale (PSS). The scale includes three sub-categories: "care and information given to the patient during treatment", "quantity and quality of treatment" and "Information and support provided to the patient and family after discharge". PSS consists of 13 items in total. Each item is scored ranging from 0 to 3 (0: Strongly disagree, 1: Disagree, 2: Agree, 3: Strongly agree). The highest score is 39 points. High scores indicate a high degree of satisfaction.
Patient satisfaction | baseline
  Patient Satisfaction from physiotherapy will be assessed Patient Satisfaction Scale in Physiotherapy (PSSP). PSSP consists of 14 items under four category subheadings of "treatment (5 items), admission (3items), logistics (4items) and global overall satisfaction (2 items)." It is a 5-point Likert type scoring scale (1 = weak, 5 = perfect). Total scores are calculated out of 100. High scores indicate a high degree of satisfaction.
Life quality | baseline
  Life quality will be assessed with SF-36 (short form). SF-36 (short form) is a general quality of life scale that evaluates physical and mental health. It consists of eight sub-dimensions and 36 items: Physical Function, Social Function, Physical Role Difficulty, Emotional Role Difficulty, Mental Health, Vitality (Energy), Pain and General Health. Scores for each subscale are calculated separately. It is scored from 0 to 100. A score of 0 from the scale indicates poor health, and a score of 100 indicates good health.

CONTACTS AND LOCATIONS:
Locations (1):
- Emel Mete, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No